CLINICAL TRIAL: NCT00388583
Title: Immunogenicity and Safety of The Split, Inactivated, Trivalent Influenza Vaccine Administered by Intradermal Route in Comparison With Intramuscular Vaccination With Standard Fluzone® in Ambulatory Elderly Subjects
Brief Title: Study of Inactivated, Split-Virion Influenza Vaccine Compared With Standard Fluzone Vaccine in Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FID04
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Orthomyxoviridae Infection; Influenza; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Inactivated Split-virion influenza vaccine; Elderly.
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — Influenza Vaccines

ARMS (2):
- Fluzone Intradermal (ID) Vaccine Group (Experimental): Participants received a dose of Fluzone Intradermal (ID) Influenza Vaccine
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine
- Fluzone Intramuscular (IM) Vaccine Group (Active Comparator): Participants received a dose of Fluzone Intramuscular (IM) Influenza Vaccine.
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Split, Inactivated, Trivalent Influenza Vaccine — 0.1 mL, Intradermal
  Other Names: Fluzone
  Arms: Fluzone Intradermal (ID) Vaccine Group
Biological: Split, Inactivated, Trivalent Influenza Vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone® 2006/2007 Formulation
  Arms: Fluzone Intramuscular (IM) Vaccine Group

SUMMARY:
As a result of the safety and immunogenicity data generated from earlier dose-ranging studies, the present formulation has been selected for further development in the elderly.

Primary Objective:

To compare the immunogenicity in subjects receiving investigational Fluzone with those of subjects receiving standard Fluzone®.

Secondary Objectives:

Immunogenicity:

To describe the immunogenicity in subjects receiving investigational Fluzone and standard Fluzone®.

Safety:

To evaluate and describe the safety profile of investigational Fluzone in terms of solicited- and unsolicited adverse events and serious adverse events post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years on the day of vaccination.
* Informed consent form signed.
* Medically stable (Subjects may have underlying illnesses such as hypertension, diabetes, ischemic heart disease, congestive cardiac disorders or hypothyroidism, as long as their symptoms/signs are controlled).
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to the standard-dose Fluzone® vaccine or a vaccine containing the same substances (the list of vaccine components is included in the Investigator's Brochure).
* Congenital or history of acquired immunodeficiency, or immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
* Systemic corticosteroid therapy as follows:
* Continuous use with a dosage equivalent to > 15 mg/day of oral prednisone for 90 days preceding vaccination
* Sporadic use with a dose of > 40 mg/day of oral prednisone for > 14 days in the 90 days preceding vaccination.

Note: Use of topical or inhalant corticosteroids is acceptable.

* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, as well as subjects who have a history of neoplastic disease and who have been disease-free for ≥ 5 years).
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures.
* Receipt of blood or blood-derived products in the past 3 months.
* Vaccination against influenza in the past 6 months.
* Any vaccination in the 4 weeks preceding the trial vaccination.
* Vaccination planned in the 4 weeks following the trial vaccination.
* Participation in another clinical trial in the 4 weeks preceding trial vaccination.
* Planned participation in another clinical trial during the present trial period. Concomitant participation in an observational trial (not involving drugs, vaccines, or medical devices) is acceptable.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Known current HIV, hepatitis B (HBsAg) or hepatitis C infection or seropositivity.
* Known thrombocytopenia or bleeding disorder contraindicating IM vaccination.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Acute illness and febrile illness with a temperature ≥ 38.0°C [or 100.4°F]) 72 hours before or on the day of inclusion.
* Received antibiotics therapy within 72 hours preceding the trial vaccination.
* Received any allergy shots in the 7-day period preceding trial vaccination and/or scheduled to receive any allergy shots in the 7-day period after trial vaccination.
* Any condition, which in the opinion of the investigator would pose a health risk to the participant.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 817 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (17):
- United States (17):
  - Alabaster, Alabama
  - Tucson, Arizona
  - Fountain Valley, California
  - Pinellas Park, Florida
  - Chicago, Illinois
  - Springfield, Missouri
  - Brooklyn, New York
  - New York, New York
  - Bensalem, Pennsylvania
  - Grove City, Pennsylvania
  - Johnstown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Fort Worth, Texas
  - Galveston, Texas
  - Layton, Utah
  - South Jordan, Utah
  - Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 28 September 2006 through 30 May 2007 in 16 clinics in the US
Pre-assignment Details: A total of 816 of the 817 participants that met the inclusion and exclusion criteria were enrolled and vaccinated. Data on the 807 participants that completed the study are presented.
Groups:
- Fluzone Intradermal (ID) Vaccine Group: Participants received a dose of Fluzone Intradermal vaccine on Day 0
- Fluzone Intramuscular (IM) Vaccine Group: Participants received a dose of Fluzone Intramuscular vaccine on Day 0
Period: Overall Study
Arm/Group | Fluzone Intradermal (ID) Vaccine Group | Fluzone Intramuscular (IM) Vaccine Group
Started | 407 | 410
Completed | 401 | 406
Not Completed | 6 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Serious Adverse Event | 2 | 0
Not completed — Did not receive vaccine | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Fluzone ID Vaccine Group: Participants received a dose (0.1 mL) of Fluzone intradermal vaccine on Day 0.
- Fluzone IM Vaccine Group: Participants received a dose (0.5 mL) of Fluzone intramuscular vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Fluzone ID Vaccine Group | Fluzone IM Vaccine Group | Total
Number analyzed (Participants) | 401 | 406 | 807
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 401 | 406 | 807
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (6.08) | 72.3 (5.83) | 72.5 (5.955)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 223 | 457
  Male | 167 | 183 | 350
Region of Enrollment [Number; unit: Participants]
  United States | 401 | 406 | 807

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least a 4-Fold Increase in Serum HAI Antibody Titer Post-vaccination With Either Fluzone Intradermal or Fluzone Intramuscular Vaccine.
Description: The serological determinations of total anti-influenza antibodies were performed using an Hemagglutinin inhibition (HAI) test.
Time Frame: Pre-vaccination and Day 28 post-vaccination
Population: Immunogenicity determination was in all per protocol population
Measure: Number; unit: Participants
Arm/Group | Fluzone Intradermal (ID) Vaccine Group | Fluzone Intramuscular (IM) Vaccine Group
Number analyzed (Participants) | 401 | 406
Participants
  A/H1N1 Serogroup (N = 400, 406) | 119 | 105 [0 to 0]
  A/H3N2 Serogroup (N = 398, 404) | 235 | 222 [0 to 0]
  B Serogroup (N = 400, 405) | 105 | 103 [0 to 0]

2. Secondary Outcome: Geometric Mean Antibody Titers (GMTs) Before and Post-vaccination With Either Fluzone Intradermal and Fluzone Intramuscular Vaccine.
Description: The serological determinations of total anti influenza antibodies were performed using an Hemagglutinin inhibition (HAI) test.
Time Frame: Pre- and Day 28 post-vaccination
Population: Immunogenicity determination was in all per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone Intradermal (ID) Vaccine Group | Fluzone Intramuscular (IM) Vaccine Group
Number analyzed (Participants) | 401 | 406
Titers
  A/H1N1 Serogroup (Pre-vaccination) | 27.46 [24.81 to 30.40] | 24.86 [22.33 to 27.69]
  A/H1N1 Serogroup (Post-vaccination) | 71.17 [63.93 to 79.22] | 59.04 [53.27 to 65.42]
  A/H3N2 Serogroup (Pre-vaccination) | 75.95 [65.42 to 88.17] | 64.95 [55.91 to 75.45]
  A/H3N2 Serogroup (Post-vaccination) | 500.65 [442.40 to 566.56] | 360.42 [317.68 to 408.91]
  B Serogroup (Pre-vaccination) | 13.11 [12.08 to 14.22] | 12.95 [11.93 to 14.05]
  B Serogroup (Post-vaccination) | 35.06 [31.91 to 38.53] | 35.77 [32.44 to 39.44]

3. Primary Outcome: Number of Participants Who Achieved Seroprotection Post-vaccination With Either Fluzone Intradermal or Fluzone Intramuscular Vaccine.
Description: Seroprotection was defined as a post-vaccination Hemagglutinin inhibition (HAI) antibody titer ≥ 40
Time Frame: Day 28 post-vaccination
Population: Immunogenicity determination was in all per protocol population
Measure: Number; unit: Participants
Arm/Group | Fluzone Intradermal (ID) Vaccine Group | Fluzone Intramuscular (IM) Vaccine Group
Number analyzed (Participants) | 401 | 406
Participants
  A/H1N1 Serogroup (N = 400, 406) | 303 | 292
  A/H3N2 Serogroup (N = 398, 405) | 391 | 389
  B Serogroup (N = 400, 406) | 200 | 213

4. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reaction, Post Vaccination With Either Fluzone Intradermal or Fluzone Intramuscular Vaccine
Description: Solicited injection site reactions: Pain, Erythema, Swelling, Induration, Ecchymosis, and Pruritus.
  Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia.
Time Frame: Day 0 up to 7 days post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants, intend-to-treat population
Measure: Number; unit: Participants
Arm/Group | Fluzone Intradermal (ID) Vaccine Group | Fluzone Intramuscular (IM) Vaccine Group
Number analyzed (Participants) | 407 | 409
Participants
  Any Injection Site Pain | 105 | 98
  Grade 3 Injection Site Pain (Incapacitating) | 0 | 1
  Any Injection Site Erythema | 282 | 49
  Grade 3 Injection Site Erythema (≥ 5 cm) | 39 | 0
  Any Injection Site Swelling | 186 | 20
  Grade 3 Injection Site Swelling (≥ 5 cm) | 17 | 4
  Any Injection Site Induration | 178 | 17
  Grade 3 Injection Site Induration (≥ 5 cm) | 12 | 0
  Any Injection Site Ecchymosis | 23 | 12
  Grade 3 Injection Site Ecchymosis (Incapacitating) | 1 | 0
  Any Injection Site Pruritus | 137 | 23
  Grade 3 Injection Site Pruritus (Incapacitating) | 0 | 0
  Any Solicited Fever | 10 | 4
  Grade 3 Solicited Fever (>102.2°F) | 0 | 1
  Any Solicited Headache | 69 | 63
  Gr 3 Solicited Headache- Prevents daily activities | 2 | 1
  Any Solicited Malaise | 57 | 41
  Grd 3 Solicited Malaise- Prevents daily activities | 3 | 4
  Any Solicited Myalgia | 68 | 56
  Grd 3 Solicited Myalgia- Prevents daily activities | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination up to 6 months post-vaccination.
Arm/Group | Fluzone Intradermal (ID) Vaccine Group | Fluzone Intramuscular (IM) Vaccine Group
Serious Adverse Events (participants affected / at risk) | 33/407 | 34/409
Other Adverse Events (participants affected / at risk) | 282/407 | 98/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fluzone Intradermal (ID) Vaccine Group (N=407) | Fluzone Intramuscular (IM) Vaccine Group (N=409)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (4) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (7) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (3) | 1 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0/0 (0)
Squamous cell carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0/0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Transuerethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device electric finding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetes mellitus non insulin dependent (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Small intestine obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fluzone Intradermal (ID) Vaccine Group (N=407) | Fluzone Intramuscular (IM) Vaccine Group (N=409)
Vessel puncture site bruise (General disorders) | 23 (23) | 15 (15)
Solicited injection site pain (General disorders) | 105/402 (105) | 98 (98)
Solicited injection site erythema (General disorders) | 282/402 (282) | 49 (49)
Solicited injection site induration (General disorders) | 178/400 (178) | 17 (17)
Solicited injection site ecchymosis (General disorders) | 23/400 (23) | 12 (12)
Solicited injection site pruritus (General disorders) | 137/402 (137) | 23 (23)
Solicited headache (Pyrexia) (Nervous system disorders) | 69/402 (69) | 63 (63)
Solicited malaise (General disorders) | 57/402 (57) | 41 (41)
Solicited myalgia (General disorders) | 68/402 (68) | 56 (56)
Solicited injection site swelling (General disorders) | 186/402 (186) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.